CLINICAL TRIAL: NCT05070013
Title: Adaptive Neurostimulation to Restore Sleep in Parkinson's Disease: An Investigation of STN LFP Biomarkers in Sleep Dysregulation and Repair
Brief Title: Adaptive Neurostimulation to Restore Sleep in Parkinson's Disease (Aim 2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0577-21-FB; 1UH3NS113769 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2021-10-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease; Sleep Fragmentation
MeSH Terms: conditions — Parkinson Disease; Sleep Deprivation | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will experience all 3 DBS stimulation interventions (one condition per week, 3 consecutive weeks): adaptive stimulation, open-loop stimulation (standard clinical stimulation therapy) and no stimulation (control). The order of stimulation conditions is randomly assigned.
Who Masked: Participant
Masking Description: To mitigate bias, participants will be blinded with respect to which stimulation intervention is assigned in each week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Adaptive Deep Brain Stimulation (Experimental): Participants will be given adaptive deep brain stimulation (DBS) during one week of at-home night sleep.
  Interventions: Device: Deep Brain Stimulation
- Open-loop Deep Brain Stimulation (Active Comparator): Participants will be given open-loop deep brain stimulation (DBS) (standard clinical stimulation therapy based on (DBS) programming for the treatment of motor symptoms) during one week of at-home night sleep.
  Interventions: Device: Deep Brain Stimulation
- No Deep Brain Stimulation (No Intervention): Deep brain stimulation (DBS) is turned off (control) during one week of at-home night sleep.

INTERVENTIONS:
Device: Deep Brain Stimulation — All participants will undergo three 1-week interventions of stimulation during nighttime sleep over the course of three consecutive weeks of in-home sleep: adaptive stimulation, open-loop stimulation and no stimulation.
  Arms: Adaptive Deep Brain Stimulation; Open-loop Deep Brain Stimulation

SUMMARY:
Parkinson's Disease (PD) is the second most common of the age-related neurodegenerative disorders, affecting over 1,900 adults per 100,000 over the age of 80 in the US. The prevalence of sleep dysfunction in PD is estimated at nearly 80-90% which includes sleep fragmentation, insomnia, rapid eye movement (REM or dream sleep) Sleep Behavior Disorder (RBD), Restless legs syndrome (RLS), periodic limb movement, excessive daytime sleepiness, and sleep apnea. Sleep is vital to homeostasis, cognition, and nervous system repair. The dysfunctional sleep accompanying PD adversely affects both motor and non-motor symptoms, resulting in diminished quality of life for both patients and caregivers, including impairments in mood and behavior, and increased morbidity and mortality. Knowledge of sleep phenomenology and pathology in humans has largely been informed by analysis of non-invasive scalp electroencephalogram (EEG), and despite the profound importance of sleep, the underlying neural circuits important for controlling sleep and wakefulness in humans remain poorly understood.

This study assesses whether adaptive stimulation of the Subthalamic Nucleus (STN) drives changes in sleep episode maintenance and improves sleep quality. Participants are adults with PD who experience inadequate motor symptom relief, and who have been offered implantation of a deep brain stimulator system targeting STN for the treatment of motor symptoms (standard-of-care). Prior to surgery, participant sleep patterns will be assessed with questionnaires and monitored with a non-invasive watch-like device. Approximately four months after implantation surgery, participants will each receive 2 1-week deep brain stimulation (DBS) treatments and 1 1-week control session with no DBS in random order. Sleep patterns will again be monitored during the treatments and compared to the patterns before surgery.

DETAILED DESCRIPTION:
IIn previous studies, investigators examined the use of local field potentials (LFP) recorded from Subthalamic Nucleus (STN) - Deep brain stimulation (DBS) electrodes to identify unique spectral patterns in STN oscillatory activity that correlate with distinct sleep cycles. This offered insight into sleep dysregulation and supported the idea that biomarkers from STN-recorded LFP could be used to identify specific sleep stages. Data from this study directly informed the development and optimization of an adaptive stimulation algorithm.

The current study will assess the efficacy of the adaptive stimulation algorithm and will test the working hypothesis that modulation of STN during nighttime sleep will normalize sleep behavior by offsetting aberrant signaling in the sleep network. Investigators will use subjective assessments, 3-week actigraphy, and nocturnal polysomnogram (PSG), in 20 Parkinson's Disease (PD) participants for 3-weeks prior to surgery and again 4-months after DBS implantation during the interventions. The time between surgery and the start of interventions allows DBS and medication to be therapeutically optimized for PD motor symptoms. Investigators will compare chronic open-loop stimulation to adaptive stimulation, and to a no-stimulation control group. All participants will experience each of the 3 interventions in random order and be blinded to the type of intervention received.

The study hopes to validate a therapeutic intervention for the burdensome non-motor symptom of sleep dysfunction in PD, and to fill a critical gap in our understanding of the contribution of STN-DBS to ameliorating sleep-wake disturbances in PD. The acquisition of these data will improve the understanding of the role of basal ganglia, specifically STN, in sleep homeostasis in PD. It is expected that STN-DBS will improve sleep-wake parameters in both the PSG and actigraphy recordings but that adaptive stimulation, targeted at sleep-stage biomarkers, will further optimize sleep and alleviate this non-motor burden in PD. Specifically, investigators predict that adaptive more so than chronic open-loop STN-DBS during sleep will decrease non-consolidated sleep, reduce the frequency of awakenings, increase the percentage time spent in REM sleep, reduce daytime sleepiness, and increase subjective experience of restfulness and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of Idiopathic Parkinson's disease (PD) with motor symptoms present for a minimum of 4 years
* Severe motor symptoms (e.g., motor fluctuations, dyskinesia, tremor, bradykinesia, rigidity) despite optimized medical therapy, that warrant surgical implantation of deep brain stimulation (DBS), according to standard clinical criteria
* Unified Parkinson's Disease Rating Scale (UPDRS-III) score off medication 20 to 80, and improvement of at least 30% in UPDRS-III score on medications, or tremor-dominant PD (score >/= 2 on UPDRS-III tremor sub-score) or tremor in addition to other motor symptoms that are treatment-resistant and result in significant functional disability
* Appropriate trials of oral PD medications resulting in inadequate relief of motor symptoms as determined by a movement disorders neurologist, and stable dose of anti-PD medications for 30 days prior to study enrollment
* Requested and approved for subthalamic nucleus deep brain stimulation surgery (STN DBS) by study site Multi-Disciplinary Movement Disorders Patient Care Conference
* Absence of abnormalities on brain magnetic resonance imaging (MRI) scan suggestive of an alternate diagnosis or serving as a contraindication to surgery
* Absence of significant cognitive deficits or significant depression (Beck Depression Inventory-II, BDI-II, score > 20) on formal Neuropsychological Testing
* Age 18 to 80 years (19 to 80 years in Nebraska)
* Able to conduct follow up neurological care exclusively at study site for duration of the RC+S INS neurostimulator device lifespan (9 years)

Exclusion Criteria:

* Any medical condition considered to elevate risk for surgical complications, such as coagulopathy,, uncontrolled hypertension, history of seizures, heart disease, inability to undergo general anesthesia, or anticoagulant medications that cannot be safely discontinued for perioperative period
* Pregnancy (women of child-bearing potential must have a negative urine pregnancy test prior to surgical procedures)
* Significant untreated depression (Beck Depression Inventory-II, BDI-II > 20 or Geriatric Depression Scale, GDS, score > 8)
* Personality or mood disorder symptoms that investigators believe will interfere with study requirements
* Required ongoing treatment with electroconvulsive therapy (ECT), repetitive transcranial magnetic stimulation (rTMS), or diathermy
* Pre-existing implanted stimulation system (e.g., cochlear implant, cardiac pacemaker, defibrillator, neuro-stimulator for indication other than Parkinson's disease), or ferromagnetic metallic implant
* Prior intracranial surgery
* History or active, drug or alcohol abuse
* Meets criteria for Parkinson's disease (PD) with Mild Cognitive Impairment (PD-MCI), as defined by Performance > 2 standard deviations below appropriate norms on tests from 2 or more of the following cognitive domains: Attention, Executive Function, Language, Memory, and Visuospatial Ability
* Restless Leg Syndrome
* Obstructive Sleep Apnea
* Inability to perform the recharge process necessary to use the RC+S brain stimulation system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency - Frequency | Baseline (days 1 - 21 before surgery) and intervention (approximately days 144 - 172)
  Sleep fragmentation frequency will be measured using FDA-approved wrist-based Actigraphy (ActiWatch Spectrum Pro). Comparisons will be made between baseline and each of the interventions.
Sleep Efficiency - Duration | Baseline (days 1 - 21 before surgery) and intervention (approximately days 144 - 172)
  Sleep fragmentation duration will be measured using FDA-approved wrist-based Actigraphy (ActiWatch Spectrum Pro). Comparisons will be made between baseline and each of the interventions.
Subjective Sleep Quality | Baseline (days 1 - 21 before surgery) and intervention (approximately days 144 - 172)
  Subjective sleep quality will be assessed using the Pittsburgh Sleep Diary. Comparisons will be made between baseline and each of the interventions.

SECONDARY OUTCOMES:
Duration of REM Sleep Stage | During intervention (approximately days 144 - 172)
  Change in the duration of rapid eye movement (REM or dream) stage sleep will be measured and compared between the 3 stimulation interventions. An artificial neural network, Dreem 3, will be used to identify sleep stage and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Abosch, MD, PhD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be available to other researchers through the Data Archive for the BRAIN Initiative (DABI) data sharing portal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting in January 2026 after the data are published.
Access Criteria: Researchers will be able to download the data after requesting access in DABI.
URL: https://dabi.loni.usc.edu